CLINICAL TRIAL: NCT01207895
Title: Molecular Determinants Affecting Fluoro-L-thymidine (FLT) Positron Emission Tomography (PET) in Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Henry C. Manning, PhD, Assistant Professor of Radiology, Neurosurgery, Biomedical Engineering, Program in Chemical and Physical Biology, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VICC GI 0993
Record Dates: First submitted 2010-09-17; First posted 2010-09-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]-FLT PET scans (Experimental)
  Interventions: Device: PET imaging with [18F]-FLT; Drug: [18F]-fluorodeoxythymidine

INTERVENTIONS:
Device: PET imaging with [18F]-FLT — Up to three [18F]-FLT PET scans; one before beginning treatment, one at week three of treatment, and one at week 11, after completion of treatment but prior to surgery.
Drug: [18F]-fluorodeoxythymidine — [18F]-fluorodeoxythymidine is administered intravenously approximately 60 minutes prior to the start of PET image acquisition.

SUMMARY:
The purpose of this study is to determine if positron emission tomography (PET) imaging with an imaging agent called 18F-fluorodeoxythymidine([18F]-FLT) will allow investigators to measure how well tumor(s) respond to treatment without taking a tissue sample (biopsy). Additionally, the investigators want to determine if it is possible to predict how well tumor(s) might respond to treatment with [18F]-FLT PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known rectal cancer.
* Subjects must have signed an approved consent form.
* Subjects must be 18 years of age or older.

Exclusion Criteria:

* Children less than 18 are excluded.
* Pregnant women and women who are breast feeding will be excluded from this study. A serum beta HCG will also be performed for each pre-menopausal female subject.
* Patients who are acutely ill who are deemed by their treating physician as not suitable candidates for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Utility of [18F]-FLT PET to assess cellular proliferation in neoadjuvant trials of patients with rectal cancer | at study entry, at week 3 during chemotherapy and radiation, and at week 11 after treatment but before surgery
  Ability of this imaging technique to determine growth of cancer cells and as a quantitative biomarker of response to relevant, molecularly targeted, therapies

SECONDARY OUTCOMES:
Correlative biology | at study entry before treatment, at week 3 of treatment, and at week 11 after treatment
  Pre-treatment and intra-treatment rectal biopsy tissue and tissue from the post-treatment surgical tumor resection will be examined for cyclin D1, TK1, PCNA, pHis-H3, thymidylate, p-Erk, p-Akt to identify changes from pre-treatment to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Manning, Ph.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/